CLINICAL TRIAL: NCT07063095
Title: Ceftazidime Plus Fosfomycin Versus Ceftazidime Alone for Severe Gram-negative Infections: a Triple-blind, Placebo-controlled Point-of-care Randomized Clinical Trial
Brief Title: A Combination Therapy With Ceftazidime and Fosfomycin Will be Compared to Ceftazidime Alone in Hospitalized Adult Patients With Suspected Severe Gram-negative Bacterial Infections
Acronym: CAVIFOS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Angela HUTTNER (Other)
Collaborators: Joint Programming Initiative on Antimicrobial Resistance (JPIAMR) (Unknown); Swiss National Science Foundation (Other)
Responsible Party: Sponsor-Investigator, Angela HUTTNER, Professor, Attending physician, Division of Infectious Diseases, University of Geneva, Switzerland
Organization: University of Geneva, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAVIFOS CCER 2024-01954
Record Dates: First submitted 2025-06-11; First posted 2025-07-14 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-08

CONDITIONS: Gram Negative Infections; Sepsis and Septic Shock
Keywords: ceftazidime; cavifos; gram-negative bacteria; intravenous fosfomycin
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — avibactam, ceftazidime drug combination; Fosfomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ceftazidime± avibactam with fosfomycin (CAZ±AVI+ FOS) (Experimental): The experimental intervention is a combination of CAZ with FOS, brand name InfectoFos®, each vial containing 2 g of fosfomycin, and 2.64 g fosfomycin disodium.
  Interventions: Drug: Ceftazidime± avibactam with fosfomycin
- Ceftazidime± avibactam with placebo (CAZ±AVI + placebo) (Placebo Comparator): Control arm will be CAZ±AVI combined with placebo.
  Interventions: Drug: Ceftazidime± avibactam with placebo

INTERVENTIONS:
Drug: Ceftazidime± avibactam with fosfomycin — The intervention will last 72h (±6h). Ceftazidime will be administered intravenously in 5% glucose serum (per hospital standard), either intermittently (divided into three doses daily) or as continuous infusion; doses will be adapted to renal function. The decision to administer CAZ by continuous infusion and to add AVI will be left to the attending physician. CAZ±AVI will be adjusted for renal insufficiency per internal guidelines of dosing and international recommendations.
  The use of CAZ with its paired beta-lactamase inhibitor avibactam, i.e., the use of ceftazidime-avibactam (Zavicefta®) instead of CAZ will occur in case of suspicion of infection by either extended-spectrum-beta-lactamase-producing Enterobacterales (ESBL-E), cephalosporinase-carrying Enterobacterales (ampC-E) or carbapenem-resistant Enterobacterales (CRE), as determined by treating physician and/or the infectious diseases consultant.
  Other Names: CAZ±AVI + FOS; InfectoFos®
  Arms: Ceftazidime± avibactam with fosfomycin (CAZ±AVI+ FOS)
Drug: Ceftazidime± avibactam with placebo — Participants randomized to the control arm will receive placebo infusion. Placebo will be 5% glucose serum and will be administered IV with the same frequency as FOS would be for the participant's renal function.
  Arms: Ceftazidime± avibactam with placebo (CAZ±AVI + placebo)

SUMMARY:
The goal of this clinical trial is to :

1. Test whether the combination of CAZ±AVI and FOS leads to superior clinical outcomes in patients with severe suspected Gram-negative bacterial infection, as demonstrated by a shorter time to normalization of quick Sequential Organ Failure Assessment (qSOFA) parameters and reduction in C-reactive protein (CRP) compared to standard of care (CAZ±AVI alone)
2. to further characterize the safety profile of this combination therapy

In the presence of such an infection, standard treatment is to start intravenous antibiotic therapy. Ceftazidime (Fortam®), or ceftazidime-avibactam (Zavicefta®), is a standard antibiotic commonly used for this purpose (for very resistant bacteria, the compound avibactam is included to protect ceftazidime from being broken down by bacteria).

Researchers will compare ceftazidime (or ceftazdime-avibactam) plus fosfomycin versus ceftazidime alone with placebo (i.e. a look-alike substance given with no drug) to examine whether the addition of another intravenous antibiotic, fosfomycin, would lead to faster recovery from severe infection and evaluate the tolerability of this combination.

Participants will:

* Be randomly assigned to either the intervention group or the control group.
* The intervention group will receive ceftazidime (with avibactam if multidrug resistant bacteria are suspected, per routine practice) and intravenous fosfomycin, and the control group will receive ceftazidime (with avibactam if multidrug resistant bacteria are suspected) and placebo.
* Either treatment will be given for 3 days, three times daily (or less frequently, depending on renal function).
* Provide a few extra blood samples (for CRP measurement, a protein marker of inflammation) during the first few days of the study.
* Be contacted in the hospital or by phone if discharged on day 28 to be asked a few questions.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥18 years)
2. Hospitalized with suspected severe Gram-negative bacterial infection
3. Signed informed consent from the patient (or oral consent from a patient with capacity but with physical inability to sign, with signed witness testimony from a person independent of the study team) of from the legal representative if the patient lacks capacity to provide informed consent

Exclusion Criteria:

1. Pregnancy or lactation
2. Known contra-indication to CAZ±AVI or FOS
3. Gram-negative directed antibiotic treatment begun >24 hours before inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Time in hours from first study-medication administration to normalization of all qSOFA parameters and decrease of peak CRP by 50%. | From date of randomization until the date of first documented normalization of qSOFA and 50% decrease in CRP. We estimate median time to be of approximately 108h and 96h in the control and intervention groups, respectively (approx 4 to 5 days)
  qSOFA scores will be collected as per routine ward practices and at minimum every 2 hours for patients with abnormal scores, until normalization.
  CRP will be measured twice daily (12 ± 4 hours apart), for 6 days or until the 50% reduction from peak is observed, whichever occurs earlier. Thereafter, measurements will be taken as clinically indicated.

SECONDARY OUTCOMES:
Incidence of adverse events of special interest (AESI) | From day 1 to day 3 (+/-1 day) of intervention and up to 48h after the last administration of the study medication/placebo
  Patients will be monitored post-randomization for the occurrence of adverse events of special interest (AESI), defined as follows:
  * New-onset pulmonary edema detected by imaging or auscultatory exam beginning during and up to 2 days after treatment with study antibiotic(s)
  * New-onset hypernatremia beginning during and up to 2 days after treatment with study antibiotic(s)
  * New-onset hypokalemia beginning during and up to 2 days after treatment with study antibiotic(s)
  * New-onset gastrointestinal events (abdominal pain, nausea, vomiting, and/or diarrhea) beginning during and up to 2 days after treatment with study antibiotic(s)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Genève, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No